CLINICAL TRIAL: NCT02312557
Title: Addition of Pembrolizumab Upon Progression on Enzalutamide in Men With mCRPC
Brief Title: Pembrolizumab in Treating Patients With Metastatic Castration Resistant Prostate Cancer Previously Treated With Enzalutamide
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Collins Medical Trust (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julie Graff, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011025; NCI-2014-02131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CR00025312; MR00044410; CRQ 2015
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2025-01-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Castration-Resistant Prostate Carcinoma; Hormone-Resistant Prostate Cancer; PSA Progression; Recurrent Prostate Carcinoma; Stage IV Prostate Adenocarcinoma Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): INITIAL TREATMENT PHASE: Patients who are progressing on enzalutamide will receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide PO daily.
  MONITORING PHASE: After completion of the initial treatment phase, patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.
  RETREATMENT PHASE: Patients with disease response or stability after the initial treatment phase will receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for an additional 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with prostate cancer that has spread to other places in the body and keeps growing even when the amount of testosterone in the body is reduced to very low levels despite previous treatment with enzalutamide. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the anti-cancer activity of pembrolizumab in men with metastatic, castration resistant prostate cancer.

SECONDARY OBJECTIVES:

I. To investigate immunological and genetic parameters to evaluate for possible markers and functional changes that are predictive of a clinical response or linked to response or resistance to PD-1 inhibition.

II. To collect circulating tumor cells (CTCs) and determine the degree to which tumor characteristics are shared by the CTCs.

III. Changes in T cell numbers, activation, and phenotype as measured in whole blood at diagnosis and throughout therapy.

IV. Systemic inflammatory markers: serum interleukin (IL)-8, IL-6, IL-1, tumor necrosis factor (TNF) and transforming growth factor (TGF)-beta.

V. Objective disease response by radiographs. VI. Prostate-specific antigen (PSA) progression free survival. VII. Overall survival. VIII. Microbiome and correlation with response.

TERTIARY OBJECTIVES:

I. Additional genetic (deoxyribonucleic acid [DNA], ribonucleic acid [RNA]) and protein analyses will be conducted to further evaluate immunotherapy and profile/characterize disease.

OUTLINE:

INITIAL TREATMENT PHASE: Patients who are progressing on enzalutamide will receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide orally (PO) daily.

MONITORING PHASE: After completion of the initial treatment phase, patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.

RETREATMENT PHASE: Patients with disease response or stability after the initial treatment phase will receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for an additional 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.

After completion of study treatment, patients are followed up at 30 days, and then every 12 weeks for 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* ENTRY CRITERIA: Metastatic, castration resistant prostate cancer progressing on enzalutamide after initial response to enzalutamide
* Histologically or cytologically confirmed adenocarcinoma of the prostate without pure small cell carcinoma; patients without histologically confirmed adenocarcinoma may be eligible if both the treating physician and the study principal investigator (PI) agree that the patient?s history is unambiguously indicative of advanced adenocarcinoma
* Be willing and able to provide written informed consent/assent for the trial
* Be >= 18 years of age on day of signing informed consent
* Have metastatic disease
* Have permission to access tissue from an archival tissue sample; (absence of archival tissue will not preclude trial participation)
* Has a metastatic deposit that can be biopsied
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL, performed within 28 days of treatment initiation
* Platelets >= 100,000/mcL, performed within 28 days of treatment initiation
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L, performed within 28 days of treatment initiation
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]); creatinine clearance should be calculated per institutional standard, performed within 28 days of treatment initiation
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN, performed within 28 days of treatment initiation
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases, performed within 28 days of treatment initiation
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (only if submitting to a biopsy), performed within 28 days of treatment initiation
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (only if submitting to a biopsy), performed within 28 days of treatment initiation
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Have a PSA or radiographic progression on enzalutamide; PSA progression is defined as two consecutive increases in PSA with the second level obtained at least 3 weeks after the first, and the second level of at least 0.5 ng/mL; soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or >= 2 new lesions on bone scan
* Have had either surgical castration OR be on luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy with serum testosterone < 50 ng/dl AND agree to stay on LHRH agonist or antagonist therapy during the study

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; the use of physiologic doses of corticosteroids may be approved after consultation with the sponsor
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier; denosumab is a prohibited medication on study and for 4 weeks prior to day 1
* Has had chemotherapy for castration-resistant disease; chemotherapy for castration-sensitive disease is permitted
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ bladder cancer that has undergone potentially curative therapy
* Has known brain metastases and/or carcinomatous meningitis
* Has a history of seizure
* Has allergy to enzalutamide
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; a severe autoimmune disease is one that requires a significant medical intervention such as hospitalization; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren?s syndrome will not be excluded from the study
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-ligand (L)1, anti-PD-L2, anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways); previous treatment with sipuleucel-T is permitted
* Has plans to receive cytotoxic chemotherapy, immune checkpoint inhibitors (eg CTLA-4 blockade), sipuleucel-T, radiopharmaceuticals, abiraterone or other experimental therapy during this study period
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has rapid progression of visceral disease and, thus is a candidate for docetaxel; this determination will be at the discretion of the treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Graff, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Graff JN, Beer TM, Alumkal JJ, Slottke RE, Redmond WL, Thomas GV, Thompson RF, Wood MA, Koguchi Y, Chen Y, Latour E, Bergan RC, Drake CG, Moran AE. A phase II single-arm study of pembrolizumab with enzalutamide in men with metastatic castration-resistant prostate cancer progressing on enzalutamide alone. J Immunother Cancer. 2020 Jul;8(2):e000642. doi: 10.1136/jitc-2020-000642. PMID 32616555

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab): INITIAL TREATMENT PHASE: Patients who are progressing on enzalutamide will receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide PO daily.
  MONITORING PHASE: After completion of the initial treatment phase, patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.
  RETREATMENT PHASE: Patients with disease response or stability after the initial treatment phase will receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for an additional 4 courses in the absence of disease progression or unacceptable toxicity. Patients continue to receive standard of care enzalutamide PO daily for the duration of the trial.
  Enzalutamide: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 58
Completed | 54
Not Completed | 4
Not completed — Survival follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 57
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: PSA Response, Defined by a PSA Decrease of at Least 50% Confirmed by a Second Measurement at Least 3 Weeks Later
Description: One-sample binomial test will be used to assess whether the proportion of PSA response (PSA decrease of at least 50%) is significantly greater than 0.05. Univariable logistic regression analysis will be conducted to assess the association between immunological parameters and PSA response responses. Scale in logit will be assessed for all continuous parameters that are identified to be significantly associated with PSA response. Descriptive statistical analysis will be conducted. The proportion estimate will be reported with 95% confidence interval.
Time Frame: Up to 30 days after completion of study treatment, up to approximately 2.5 years total.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 58
Participants | 11
Statistical Analysis 1: Comparison: Treatment (Pembrolizumab); Test type: Other; p < 0.01, One-sample binomial test of proportion; Proportion = 0.19, 95% CI 2-sided [0.09 to 0.29]

2. Secondary Outcome: Changes in T Cell Activation as Measured in Whole Blood
Description: Descriptive statistical analysis will be conducted. The proportion estimate will be reported with 95% confidence interval, and the continuous variables will be summarized using nmissing, mean, std, median, min, and max.
Time Frame: Baseline to up to 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Changes in T Cell Numbers as Measured in Whole Blood
Description: as for outcome 2
Time Frame: Baseline to up to 4 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Changes in T Cell Phenotype as Measured in Whole Blood
Description: as for outcome 2
Time Frame: Baseline to up to 4 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Circulating Tumor Cells
Description: as for outcome 2
Time Frame: Up to 4 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Deoxyribonucleic Acid Mutation
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

7. Secondary Outcome: Immunohistochemistry for PD-1, PD-L1 and PD-L2 in Prostate Tissue
Description: as for outcome 2
Time Frame: Baseline
Reporting Status: Not Posted

8. Secondary Outcome: Immunological Parameters, Including Leukocytes, Lymphocytes, and Macrophages in Prostate Tissue
Description: as for outcome 2
Time Frame: Baseline
Reporting Status: Not Posted

9. Secondary Outcome: Objective Disease Response by Radiographs
Description: Descriptive statistical analysis will be conducted. The proportion estimate will be reported with 95% confidence interval.
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

10. Secondary Outcome: Overall Survival
Time Frame: Up to 2.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 58
months | 17.6 [14.7 to 23.0]

11. Secondary Outcome: Percent Change in PSA
Description: Descriptive statistical analysis will be conducted. The proportion estimate will be reported with 95% confidence interval, and the continuous variables will be summarized using number (n)missing, mean, standard deviation (std), median, minimum (min), and maximum (max).
Time Frame: Baseline to up to 30 days after completion of study treatment
Reporting Status: Not Posted

12. Secondary Outcome: PSA Progression Free Survival, Where the Definition of Progression Will be PSA Progression Per Prostate Cancer Working Group 2 Criteria
Description: If there is a decline from baseline, progression is an increase in PSA that is 25% and 2 ng/ml above the nadir, which is confirmed by a second value 3 or more weeks later (i.e., a confirmed rising trend). Kaplan-Meier curve will be plotted to illustrate the PSA progression free survival for all, and for subgroups (abiraterone versus no prior abiraterone and sipuleucel-T versus no prior sipuleucel-T).
Time Frame: Up to 2.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 58
months | 4.3 [3.4 to 7.6]

13. Secondary Outcome: Systemic Inflammatory Markers (Serum IL-8, IL-6, IL-1, TNF and TGF-beta)
Description: as for outcome 2
Time Frame: Up to 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: After the end of treatment, each subject will be followed for 30 days for adverse event monitoring. Serious adverse events will be collected for 90 days after the end of treatment. If the investigator learns of any AEs or SAEs related to pembrolizumab beyond the 90 days but less than 2.5 years, then that will be captured.
Description: The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 4.0.
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 3/58
Serious Adverse Events (participants affected / at risk) | 27/58
Other Adverse Events (participants affected / at risk) | 55/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=58)
Myelitis (Nervous system disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Diabetes mellitus I (Endocrine disorders) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary tract infection (Infections and infestations) | 1
Hematuria (Renal and urinary disorders) | 3
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Enterocolitis infectious (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Fall (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 2
Pain (General disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anemia (Investigations) | 1
Hypercalcemia (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=58)
Fatigue (General disorders) | 13
Diarrhea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 11
Palpitations (Cardiac disorders) | 2
Pain (General disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 9
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Hypertension (Vascular disorders) | 26
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 6
Anemia (Blood and lymphatic system disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 13
Urinary incontinence (Renal and urinary disorders) | 3
Fecal incontinence (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 4
Constipation (Gastrointestinal disorders) | 11
Urinary tract obstruction (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Bladder spasm (Renal and urinary disorders) | 2
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 7
Weight loss (Investigations) | 5
Dizziness (Nervous system disorders) | 6
Dry mouth (Gastrointestinal disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Mass on arm (Musculoskeletal and connective tissue disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Myelitis (Nervous system disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Upper respiratory infection (Infections and infestations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 3
Amnesia (Nervous system disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Fungal infection (Infections and infestations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 3
Facial nerve disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Watering eyes (Eye disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 5
Alanine amonitransferase increased (Investigations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Endocrine disorders other, sweats (Endocrine disorders) | 1
Edema limbs (General disorders) | 3
Floaters (Eye disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Platelet count decreased (Investigations) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Diabetes mellitus 1 (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Penile infection (Infections and infestations) | 1
Conjunctivitis (Eye disorders) | 1
Headache (Nervous system disorders) | 1
Radiculitis (Nervous system disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cataract (Eye disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Stye (Eye disorders) | 1
Pain (General disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Skin and subcutaneous tissue disorders - red patch left cheek (Skin and subcutaneous tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Skin and subcutaneous tissue disorders - cut, right forearm (Skin and subcutaneous tissue disorders) | 1
Memory impairment (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hot flashes (Vascular disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pain, shoulder (Musculoskeletal and connective tissue disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Tachycardia (Cardiac disorders) | 1
Tremor (Nervous system disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Chills (General disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Weight gain (Investigations) | 1
Dysgeusia (Nervous system disorders) | 2
Skin induration (Skin and subcutaneous tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Localized edema (General disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2
Renal calculi (Renal and urinary disorders) | 1
Tooth infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Glaucoma (Eye disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
CPK increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT02312557/Prot_SAP_000.pdf